CLINICAL TRIAL: NCT00450593
Title: Studies of Familial Melanoma
Brief Title: Identifying Gene Mutations in Patients With Melanoma and in Families With a History of Hereditary Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-LCC-99/3/45; CDR0000532941 (Registry Identifier: PDQ (Physician Data Query)); EU-20705
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Hereditary Multiple Melanoma; Melanoma (Skin)
Keywords: melanoma; hereditary multiple melanoma; recurrent melanoma; stage 0 melanoma; stage IV melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma, Cutaneous Malignant; Melanoma | interventions — Gene Expression Profiling; Microarray Analysis; Genetic Testing

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: molecular genetic technique
Genetic: mutation analysis
Other: laboratory biomarker analysis
Procedure: mutation carrier screening
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Identifying gene mutations and other risk factors in patients with melanoma and in families with a history of hereditary melanoma may help doctors identify persons at risk for melanoma and other types of cancer. It may also help the study of cancer in the future.

PURPOSE: This clinical trial is studying gene mutations in patients with melanoma and in families with a history of hereditary melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence and etiologic significance of variants of known melanoma susceptibility genes (MSGs) in families with multiple cases of melanoma.
* Determine the proportion of multiple-case families that are explained by high-penetrance mutations in known MSGs.
* Determine the proportion of multiple-case families that are explained by these mutations and whether it varies with latitude, as a surrogate for ultraviolet exposure, with number of affected relatives, with average age at onset of melanoma in relatives, with presence of multiple primary melanoma, or with other family-specific variables.
* Determine the penetrance of MSG mutations in these families.
* Determine if the penetrance varies with age, sex, or birth cohort.
* Determine if the penetrance varies with the gene involved or nature of the mutation.
* Assess the penetrance in mutations that also have a deleterious effect on the alternative splice product, p14ARF.
* Determine whether carriers of MSGs have an increased susceptibility to other types of cancer.
* Determine the risk of other types of cancers for mutation carriers.
* Determine environmental exposures, in particular sun exposure, that modify risk of melanoma in MSG mutation carriers.
* Determine the cutaneous phenotypes that correlate with melanoma risk in these families.
* Correlate cutaneous phenotypes with the presence of MSG variants.
* Determine the effect of other covariates, such as sun exposure or the presence of alleles of putative modifying genes (e.g., MC1R or CDKN2A), on phenotype.
* Determine if modifier genes, such as those controlling pigmentation of the skin, and therefore sun susceptibility, modify risk in MSG mutation carriers.
* Identify any histopathological correlates of MSG status in primary tumors arising in melanoma-susceptible individuals in these families.
* Identify any histopathological correlates of primary melanomas in carriers of MSG mutations with other covariates.

OUTLINE: This is a case-control, multicenter study.

Participants complete 2 questionnaires and assist in the creation and expansion of a family pedigree. Blood samples are examined for melanoma susceptibility gene mutations, including CDK4 and CDKN2A.

Participants are also examined for moles and photographed. Physical variables (e.g., skin, eye, and hair pigmentation) and sun damage (solar lentigines and freckling) are also noted.

If available, tissue samples are examined for Clark level, Breslow thickness, and frequency of mitoses. Peri-lesional skin from tumors is examined by p53 staining.

Participants are followed periodically to monitor cancer development.

Peer reviewed and funded or endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 5,000 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Prior multiple primary melanomas

    * Histological samples available
  * Family history of melanoma, with melanoma in two first-degree relatives (e.g., cases of melanoma in both a mother and son or in two brothers but not in two cousins)
  * Family history of melanoma, where three or more individuals (of any relationship) have had melanoma

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 1989-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Predictive significance of melanoma susceptibility gene (MSG) mutations in the CDKN2A gene
Susceptibility to other types of cancer as a feature of MSG mutations
Risk of other types of cancers in mutation carriers
Environmental exposures, in particular sun exposure, that modify risk of melanoma in MSG mutation carriers

CONTACTS AND LOCATIONS:
Overall Officials: Julia Newton Bishop, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom